CLINICAL TRIAL: NCT03231527
Title: Multicentric Registry Database of Total Arterial CABG
Brief Title: Outcomes of Total Arterial Coronary Artery Bypass Grafting
Acronym: MOZART
Status: Withdrawn | Type: Observational
Why Stopped: research group's decision
Sponsor: University of Glasgow (Other)
Collaborators: Campus Bio-Medico University (Other); Universitaire Ziekenhuizen KU Leuven (Other); Thorax Centrum Twente (Other); Golden Jubilee National Hospital (Other Government)
Responsible Party: Principal Investigator, Cristiano Spadaccio, Cardiothoracic surgeon, University of Glasgow
Other Study IDs: UG-002
Record Dates: First submitted 2017-07-24; First posted 2017-07-27 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: Coronary Artery Disease; Surgical Wound Infection
MeSH Terms: conditions — Coronary Artery Disease; Surgical Wound Infection | interventions — Coronary Artery Bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Total Arterial coronary CABG: Total Arterial revascularization
  Interventions: Procedure: coronary artery bypass grafting (CABG)
- Saphenous vein based CABG: Saphenous vein based revascularization
  Interventions: Procedure: coronary artery bypass grafting (CABG)

INTERVENTIONS:
Procedure: coronary artery bypass grafting (CABG) — myocardial revascularization

SUMMARY:
"real-life" retrospective multicentric database for the analysis of the long term outcomes of total arterial CABG in comparison to saphenous vein based CABG

DETAILED DESCRIPTION:
This aim of this registry is to create a multi centric database for the analysis of basic long term outcomes and immediate postoperative outcomes of total arterial CABG in comparison to saphenous vein based CABG. The registry will include both on pump and off pump surgery. The registry is intended to capture the "real-life" picture of the CABG scenario among centers worldwide

ELIGIBILITY:
Inclusion Criteria:

* elective CABG patients (on pump or off pump surgery; pedicles of skletonized internal mammary artery harvesting technique; open or endoscopic vein harvesting technique)

Exclusion Criteria:

* urgent or emergent CABG
* concomitant procedures
* redo cases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary elective isolated CABG from multivessel coronary artery disease (CAD
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-11 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Survival | data collection every year up to 5 years after operation/entry in the registry
  Long term survival
MACCEs | data collection every year up to 5 years after operation/entry in the registry
  Major cardiac events (myocardial infarction, stroke, readmission for CHF)
target vessel revascularization | data collection every year up to 5 years after operation/entry in the registry
  readmission for revascularization due to graft failure
Wound infection | data collection every year up to 5 years after operation/entry in the registry
  Readmission for wound infection (superficial sternal wound infection, deep sternal wound infection, saphenous vein related wound infection, need for VAC therapy, need for surgical debridment, need for prolonged antibiotic therapy)

SECONDARY OUTCOMES:
Blood product usage | perioperative (in hospital)
  unit of concentrated red cells, fresh frozen plasma, platelets
Bleeding | perioperative (in hospital)
  surgical bleeding requiring re-exploration
Length of ICU stay | perioperative (in hospital)
  number of days in ICU
Length of hospital stay | perioperative (in hospital)
  number of days in hospital
Duration of ventilation | perioperative (in hospital)
  number of hours ventilated
Cardiac complication | perioperative (in hospital)
  prolonged inotropic support (more than 48 hrs), IABP, ECMO
Respiratory complications | perioperative (in hospital)
  pneumonia, reintubation, pneumothorax requiring drainage, effusion requiring drainage
Renal complications | perioperative (in hospital)
  acute kidney injury not requiring dyalisis, dialysis
GI complications | perioperative (in hospital)
  mesenteric ischemia requiring surgery, ileus

CONTACTS AND LOCATIONS:
Overall Officials: Cristiano Spadaccio, MD, PhD, Principal Investigator — Golden Jubilee National Hospital
Locations (4):
- Campus St Ian, Genk, Belgium
- University Campus Bio-Medico, Rome, Italy
- Thoracic Centrum Twente, Enschede, Netherlands
- Golden Jubilee National Hospital, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No